CLINICAL TRIAL: NCT06230549
Title: Prospective Randomized Validation of Adaptive Radiotherapy in Patients With Gynecological Tumors and Indication for Radiotherapy
Brief Title: Adaptive Radiotherapy in Patients With Gynecological Tumors
Acronym: ProART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Maja Guberina, PD Dr. med. (MD) M. Guberina (senior consultant, specialist), University Hospital, Essen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 23-11675-BO
Record Dates: First submitted 2023-12-30; First posted 2024-01-30 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Gynecological Tumor; Adaptive Radiotherapy; Radiation; Curative Treatment; Optimization; Adaptive Radiation Therapy; Image Guided Radiotherapy; Cervical Carcinoma
Keywords: gynecological tumor; adaptive radiotherapy; radiation; curative treatment; optimization; adaptive radiation therapy; image guided radiotherapy; Cervical carcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Interventional Arm (Experimental): Adaptive Radiotherapy
  Interventions: Radiation: Adaptive Radiotherapy
- Standard conventional Treatment Arm, IGRT (Active Comparator): Standard conventional Treatment Arm, IGRT
  Interventions: Radiation: Adaptive Radiotherapy

INTERVENTIONS:
Radiation: Adaptive Radiotherapy — Adaptive Radiotherapy, online onboard adaptation of dose distribution with a specialist radiation oncologist and a medical physicist
  Other Names: Adaptive Radiation Therapy

SUMMARY:
Prospective randomized evaluation of adaptive radiotherapy in the definitive radiotherapy of locally advanced gynecologic carcinoma (e.g. cervical carcinoma, endometrial carcinoma, vaginal carcinoma), in the postoperative situation or first series of external beam radiotherapy and in patients in whom radical surgery or HDR brachytherapy as dose boost is not an option.

DETAILED DESCRIPTION:
Online-adaptive radiotherapy (ART) makes it possible to adapt the dose distribution to the anatomical changes online immediately before each radiation fraction. Adaptive radiotherapy is a further development of image-guided radiotherapy (IGRT), which is now standard in radiotherapy. Here, a cone-beam CT (CBCT) is also performed at the beginning of each fraction, which is used to position the patients in relation to the radiation field arrangement of the initial radiation plan approved for the series. In contrast to ART, with IGRT the radiation plan cannot be adapted to deformations in the body from radiation fraction to radiation fraction, e.g. due to different rectum and bladder fillings.

In ART mode, the online adaptive treatment plan for the current treatment is then selected and approved by the specialist online onboard in all cases in which the current target volume for the tumor expansion is not sufficiently covered by the initial treatment plan pre-planned for the series with its planned tolerances, or surrounding normal tissue is exposed too much. If the ART plan does not show any clear dosimetric advantages over the reference plan, especially if the initial plan covers the target volume of the day well, there are no dose increases and the normal tissues are spared as intended, the initial radiation plan from the planning CT can also be used as in IGRT. The aim of this study is to treat at least 15 patients with locally advanced gynecological carcinoma (mainly cervical carcinoma, endometrial carcinoma, vaginal carcinoma), who are to receive definitive radiotherapy at the Department for Radiotherapy at the University Hospital Essen, in ART mode on the Ethos therapy device over an initial 10 radiation fractions. The dose distribution is always compared with the adaptive and the initial plan for the radiation series on the anatomy of the day by the specialist and medical physics expert. The aim of this study is to prospectively investigate what percentage of patients benefit from ART when using standard PTV margins and how to recognize the corresponding patients early in the series. Secondarily, it will be investigated in what proportion of patients the risk organ burden and the safety margins around the clinical target volume can be reduced with ART compared to IGRT and how large this reduction can be.

The EORTC and CTC AE toxicitiy scales and further assessment scales will be evaluated in order to quantify objective and subjective side effects.

ELIGIBILITY:
Inclusion Criteria:

ECOG 0-1 confirmation by histophatology MR of the pelvis staging

Exclusion Criteria:

Recurrent disease Prior Radiotherapy in pelvic region stage pM1 or cM1

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2026-12-15 (Estimated)

PRIMARY OUTCOMES:
Rectal Toxicity | 2 weeks to 5 years
  Rectum, EORTC CTC-AE (Common Toxicity Criteria (CTC) of the European Organisation for Research and Treatment of Cancer (EORTC)) 1-5, [score 1: nearly no toxicity, asymptomatic changes - score 5: worst outcome (death)]
Bladder Toxicity | 2 weeks to 5 years
  Bladder, EORTC CTC-AE (Common Toxicity Criteria (CTC) of the European Organisation for Research and Treatment of Cancer (EORTC)) 1-5, [score 1: nearly no toxicity, asymptomatic changes - score 5: worst outcome (death)]
Skin Toxicity | 2 weeks to 5 years
  Skin, EORTC CTC-AE (Common Toxicity Criteria (CTC) of the European Organisation for Research and Treatment of Cancer (EORTC)) 1-5, [score 1: nearly no toxicity, asymptomatic changes - score 5: worst outcome (death)]
Lymph-Edema grade | 2 weeks to 5 years
  Lymph-Edema, EORTC CTC-AE ( (Common Toxicity Criteria (CTC) of the European Organisation for Research and Treatment of Cancer (EORTC)) 1-3, [score 1: nearly no toxicity, asymptomatic changes - score 3: worst outcome, severe symptoms; limiting self care ADL]

SECONDARY OUTCOMES:
Overall Survival | 5 years
  Overall Survival
Progression Free Survival | 5 years
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Department for Radiotherapy, University Hospital Essen, National Center for Tumor Diseases (NCT) West, Essen, Germany / NRW, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guberina M, Santiago Garcia A, Khouya A, Pottgen C, Holubyev K, Ringbaek TP, Lachmuth M, Alberti Y, Hoffmann C, Hlouschek J, Gauler T, Lubcke W, Indenkampen F, Stuschke M, Guberina N. Comparison of Online-Onboard Adaptive Intensity-Modulated Radiation Therapy or Volumetric-Modulated Arc Radiotherapy With Image-Guided Radiotherapy for Patients With Gynecologic Tumors in Dependence on Fractionation and the Planning Target Volume Margin. JAMA Netw Open. 2023 Mar 1;6(3):e234066. doi: 10.1001/jamanetworkopen.2023.4066. PMID 36947038